CLINICAL TRIAL: NCT04960254
Title: Prevalence of Internet Gaming Addiction in Adolescent
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, lecturer, resarcher OF Neurology and Psychiatry department, Assiut University
Other Study IDs: internet gaming addiction
Record Dates: First submitted 2021-03-30; First posted 2021-07-13 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Addictive Behavior; Adolescent Behavior
MeSH Terms: conditions — Behavior, Addictive; Adolescent Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: internet gaming addiction — The Strengths and Difficulties Questionnaire (SDQ) parent : to asses behavioural change Socioeconomic Scale:It contains four main variables:1-The educational level of the father and mother.2-The occupation of the father and mother. 3-Total family income. 4-life style of the family.
  Emotional Avoidance Strategy Inventory for Adolescents (EASI):The EASIA is a 17-item (Kennedy & Ehrenreich-May 2017) measure assessing the use of emotionally avoidant strategies in adolescents.
  The internet gaming addiction scale : t is used to evaluate internet gaming addiction.

SUMMARY:
Excessive problematic use of the internet has been a topic of discussion in the academic literature for many years and has gained more attention recently. The majority of those at risk are in early adulthood. Pathological internet use (PIU) is also termed internet addiction disorder (IAD), with both terms used to link internet use with addiction terminology.

Consistent with other psychiatric conditions such as depression symptoms, PIU prevalence rates among adolescents vary widely from as low as 0.3% to 38%. Likewise, PIU prevalence among college students (young adults) showed a wide variation ranging from 3% to 34%, worldwide. Nowadays, internet gaming addiction became a problematic issue in adolescent.

This is a case -control study, aimed to evaluate the prevalence and risk factors of internet gaming addiction among adolescents and its relationship with emotion regulation and comorbid psychiatric disorders.

ELIGIBILITY:
Inclusion criteria:

1. Both males and females were included.
2. Age ranges from 10- 18 years.
3. Willing of the parents or the caregivers to participate in the study.

Exclusion criteria:

* Children with intelligence quotient below 70.
* Children with history of substance use or psychiatric disorders.
* Children with medical or other neurological conditions.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Egyptian adolescent will be the target population. Target students will be selected randomly by using a multistage stratified cluster sampling technique.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-12-06 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
measure prevalence of internet gaming addiction in adolescent | through study completion, an average of 1 year
  by using internet gaming addiction scale that a cut-off of 32 was adequate to distinguish between disordered and non-disordered gamers
measure possible risk factor of internet gaming addiction in adolescent | through study completion, an average of 1 year
  by using the Strengths and Difficulties Questionnaire (SDQ) that higher score will be more disturbed

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdel-Salam DM, Alrowaili HI, Albedaiwi HK, Alessa AI, Alfayyadh HA. Prevalence of Internet addiction and its associated factors among female students at Jouf University, Saudi Arabia. J Egypt Public Health Assoc. 2019 Feb 26;94(1):12. doi: 10.1186/s42506-019-0009-6. PMID 32813134
- [Result] Ahmer Z, Tanzil S. Internet addiction among social networking sites users: Emerging mental health concern among medical undergraduates of Karachi. Pak J Med Sci. 2018 Nov-Dec;34(6):1473-1477. doi: 10.12669/pjms.346.15809. PMID 30559806